CLINICAL TRIAL: NCT07147478
Title: Video Analysis and Artificial Intelligence for the Analysis of Upper Limb Movement in Children. Validation of a Technique in a Pediatric Population Aged 6 to 17 Years
Brief Title: Video Analysis and Artificial Intelligence for the Analysis of Upper Limb Movement in Children
Acronym: AIME
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240471; IDRCB 2024-A00896-41 (Other: ANSM)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Clinical Examination of the Shoulder; Video-assisted Clinical Examination
Keywords: Clinical Examination of the Shoulder; Video-assisted clinical examination; Artificial intelligence; ShoulderLoc; Goniometer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
The principle of the study is to compare the data obtained using a shoulder movement analysis software with those obtained during a traditional clinical examination, that is, using a goniometer and the modified Mallet classification

DETAILED DESCRIPTION:
The children are recorded performing 3 sets of shoulder movements (abduction, adduction, flexion, extension, external rotation 1, external rotation 2, internal rotation 2), first on the left and then on the right, at maximum active range of motion, chosen active range of motion, and maximum passive range of motion. The recordings are made by an RGB-D camera connected to a software (ShoulderLoc from B-com) equipped with artificial intelligence that, after image processing, determines the joint range angle of the shoulder for the given movement. This value is compared to the visual estimation of the examiner and its measurement using a goniometer. The hand-mouth, hand-neck, and internal rotation 1 movements are also performed and compared with the data from the modified Mallet classification.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 17 years old at the time of inclusion
* No neurological pathology
* No history of upper limb surgery
* No upper limb trauma above the hand in the 6 months preceding the examination
* Ability to stand for a minimum of 2 minutes
* Consent from the child, both parents, and/or legal representatives for participation in a filmed clinical examination.

Exclusion Criteria:

* Inability to understand the different movements requested.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from the orthopedic and trauma consultation or the orthopedic hospitalization department, aged 6 to 17, without any upper limb disorders.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of a video-assisted clinical examination method with commonly used clinical practices | 1 day
  Perform 2 sets of 7 to 10 shoulder movements, both active and passive, measure mobility angles using a goniometer and the Mallet classification, as well as the ShoulderLoc software and its artificial intelligence program. Compare the averages obtained for each movement using both methods and compare them using an intraclass correlation coefficient (ICC).

SECONDARY OUTCOMES:
Measurement of optimal acquisition distances for video quality, | 1 day
  Validate the methodology and protocol for acquiring video movements in children
Exam duration based on age | 1 day
  Validate the methodology and protocol for acquiring video movements in children
Technical difficulties. | 1 day
  Validate the methodology and protocol for acquiring video movements in children
Obtain objective, quantified data on pure and combined shoulder movements | 1 day
  Description of results obtained by video recording a series of successive movements and analyzing them with artificial intelligence that allows for angle calculations.
Compare measurements obtained in active and passive motion for the same movement, through video measurement and manual (goniometer) measurement, to simple visual estimation measurements. | 1 day
  Comparison of the average angles obtained in active and passive motion using different methods, compared to visual assessment.
Study the satisfaction of the contribution of video tools in daily clinical practice | 1 day
  Data collection to assess feasibility in daily clinical practice (subgroup studies concerning equipment usage parameters to propose a protocol adapted to children's age).

CONTACTS AND LOCATIONS:
Overall Officials: Manon BACHY-RAZZOUK, MCU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Chirurgie Orthopédique et Réparatrice de l'Enfant - Hôpital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No